CLINICAL TRIAL: NCT01085240
Title: Getting on With the Rest of Your Life After Stroke: A Cross-Canada Program Aimed at Enhanced Life Participation, Prevention of Deterioration and Optimization of Health Care Utilization
Brief Title: Getting on With the Rest of Your Life After a Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Canadian Stroke Network (Other)
Responsible Party: Principal Investigator, Nancy Mayo, PhD, McGill University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: A12-B44-06A
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Start Later (Other): The participants receive the Mission Possible intervention but it is delayed by 3 months.
  Interventions: Other: Mission Possible
- Start Now (Experimental): The participants start the Mission Possible program right away.
  Interventions: Other: Mission Possible

INTERVENTIONS:
Other: Mission Possible — The intervention focuses on leisure education, exercise and community re-integration.
  Other Names: Participation

SUMMARY:
The primary objective is to determine the extent to which participation in life's roles can be optimized through the provision of a community-based structured program providing the opportunity for physical activity, leisure, and social interaction.

A secondary objective is to estimate the extent to which participation is associated with health benefits including health-related quality of life and reduction of unplanned health-care encounters for the person with stroke and reduction of burden and improvement in quality of life for caregivers.

DETAILED DESCRIPTION:
In the fall of 2004, a group of rehabilitation researchers developed a protocol for a cross-Canada randomized trial aimed at enhancing life participation after stroke. This project was an important part of the CSN's program and its renewal submission to the Networks of Centers of Excellence. In December 2004 the Canadian Stroke Network agreed to fund pilot work for this ambitious project, spread over six sites. The pilot funding permitted key aspects of the protocol to be developed and put in place: (i) elements of the intervention have been chosen (physical activity, leisure and social) (ii) the assessment tools have been chosen and tested; (iii) community-based partner organizations have been identified; and (iv) the intervention prototype has been tested for feasibility.

The primary objective of the main trial is to determine the extent to which participation in life's roles can be optimized through the provision of a community-based structured program providing the opportunity for physical activity, leisure, and social interaction. A secondary objective is to estimate the extent to which participation is associated with health benefits including health-related quality of life and reduction of unplanned health-care encounters for the person with stroke and reduction of burden and improvement in quality of life for caregivers. In this context, the meaning of "participation" is as defined by the World' Health Organization (WHO) and reflects both society's and the person's perspective.

The target population will be persons living in the community who have completed all formal institution-based, in-patient and ambulatory, rehabilitative interventions. No restriction on time since stroke will be imposed. Excluded will be persons who are already enrolled in existing community based projects and persons with cognitive impairment.

Sites: Six sites participated in the feasibility phase. Information emanating from these sites as well as dissemination activities of the CSN and the Canadian Stroke Strategy, have led to interest expressed by other sites across Canada prepared to run the trial phase of this project.

The study design proposed is a two-period, site-stratified, randomized, crossover design with timing of entry randomized to immediate entry or delayed entry so that there is about a six month time difference between groups. The intervention period is 9 months and the follow-up period is an additional 6 months (total 15 mos.) This design would provide for both assessment of between- group and within-person change. The main outcome is the amount of time spent in meaningful activity during the day (outcome related to primary objective).

Sample size required to have sufficient power to detect between-group differences is 240 subjects from sites across Canada. As there is considerable interest in community reintegration, "snowball" entry of sites would make it more realistic to accumulate sample size and would also make the results more generalizable and locally responsive.

ELIGIBILITY:
Inclusion Criteria:

* living in the community
* who have completed all formal institution-based, in-patient and ambulatory, rehabilitative interventions.

Exclusion Criteria:

* already enrolled in existing community based projects
* persons with cognitive impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Participation | baseline, 3, 6, 12 and 15 months
  participation in leisure measured using the CHAMPS

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Mayo, PhD, Principal Investigator — Division of Clinical Epidemiology
Locations (1):
- Division fo Clinical epidemiology, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082